CLINICAL TRIAL: NCT00826527
Title: Evaluation of Solifenacin in the Treatment of OAB Symptoms in Patients Who Have Successfully Undergone GreenLight Photoselective Vaporization of the Prostate (PVP)for the Treatment of Clinically Significant Benign Prostate Hyperplasia (BPH)
Brief Title: Evaluation of Solifenacin in the Treatment of OAB Symptoms in Patients Who Have Successfully Undergone GreenLight Photoselective Vaporization of the Prostate (PVP)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Urology Research Center (Other)
Responsible Party: Jeffrey M. Frankel, MD, Seattle Urology Research Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SURC-01-2006
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Urinary Frequency; Urinary Urgency; Nocturia
MeSH Terms: conditions — Nocturia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Solifenacin PO — Tab 5 mg Daily for 12 Weeks

SUMMARY:
The purpose of this study is to demonstrate that solifenacin post-operatively improves irritative symptoms in men whose obstructive symptoms have been relieved with the GreenLight laser outpatient procedure.

DETAILED DESCRIPTION:
Obstruction of the urinary tract secondary to benign prostatic hyperplasia can result in both obstructive and irritative urinary symptoms. In the last few years, photovaporization of the prostate has emerged as a popular teatment for this problem. This outpatient procedure uses a GeenLight KTP laser manufactured by Laserscope to vaporize the obstructing aspects of the prostatic urethral tissue to create a central cavity. After obstruction is relieved , it is not uncommon for a patient to be left with the irritative symptoms of frequency, urgency and nocturia, either from the procedure itself in the short-term or due to changes that develop in the bladder due to the long-standing obstruction. Clinical experience with this procedure indicates that after the mechanical obstruction of the prostate is relieved, medical therapy with an antimuscarinic agent should be able to alleviate these irritative urinary symptoms without the risk of urinary retention. By adding solifenacin in the early post operative period ( 2-12 weeks)for the subset of patients still experiencing irritative symptoms, further improvements in bladder symptoms my be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Male patients greater than 18 years of age with continued OAB symptoms after successful PVP for BPH.
* Patients may be included if they have previously been treated with FDA approved anticholinergic agents for the treatment of OAB such as Oxybutynin chloride(generic oxybutynin chloride, Ditropan XL, or Oxytrol) Tolterodine tartrate(Detrol or Detrol LA), or trospium chloride(Santura) and are no longer receiving such treatment for a minimun of 14 days prior to study

Exclusion Criteria:

* Previous treatment with darifenacin
* Urinary obstruction as defined as a Qmax < 12 ml/sec at time of study entry.
* Urinary retention as defined as PVR > 150 ml
* Neurogenic Bladder
* Prostate Cancer
* Chronic inflammation( i.e. interstitial cystitis)
* Bladder stones
* History of bladder cancer
* Urinary tract infection
* Uncontrolled narrow-angle glaucoma
* Gastric retention
* History of diagnosed gastro-intestinal obstructive disease.
* Severe renal or hepatic impairment
* Concomitant anticholinergic or antispasmodic medications.
* Known or suspected hypersensitivity to Solifenacin, any of its components (lactose monohydrate, corn starch, hydromellose 2910, magnesium stearate, talc, polyethylene glycol 8000 ant titanium dioxide with yellow ferric oxide(5 mg tablet) or red ferric oxide(10 mg tablet, or other anticholinergics.
* Participation in any clinical trial involving an investigational drug, within 30 days prior to enrollment.
* Any clinical condition, which in the opinion of the investigator, would not allow safe completion of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of micturitions per 24 hours utilizing a 3 day micturition diary | 12 weeks

SECONDARY OUTCOMES:
Change in mean nocturia episodes/24 hours based on 3 day diary | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M Frankel, MD, Principal Investigator — Seattle Urology Research Center
Locations (1):
- Seattle Urology Research Center, Seattle, Washington, United States